CLINICAL TRIAL: NCT02180035
Title: Effect of Treatment Nutritional With Supplementation About Biochemical Profile and Anthropometry in Adult Patients With HIV/AIDS
Brief Title: Treatment With Nutritional Eating Plan and Dietary Fibers in Adult Patients With HIV/AIDS
Acronym: PRECOR-NUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Marianne de Oliveira Falco, Effect of Treatment With Nutritional Eating Plan and Supplementation With Dietary Fibers in Adult Patients With HIV / AIDS, Conselho Nacional de Desenvolvimento Científico e Tecnológico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNPq- 478741/2008-1
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Dietary Modification; Dyslipidemia; Signs and Symptoms, Digestive; HIV
Keywords: diet therapy; symbiotic; dyslipidemia; gastrointestinal symptoms; body composition; adherence; HIV; HAART
MeSH Terms: conditions — Dyslipidemias; Signs and Symptoms, Digestive | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Symbiotic & Nutritional intervention (Experimental): Symbiotic (dietary fibers + probiotic bacteria) 6g sachet twice daily for 6 months, dietary prescription and nutritional counseling
  Interventions: Dietary Supplement: Symbiotic; Behavioral: Nutritional intervention
- Maltodextrin & Nutritional intervention (Placebo Comparator): Maltodextrin (placebo for symbiotic) 6g sachet twice daily for 6 months, dietary intervention and nutritional counseling.
  Interventions: Dietary Supplement: Maltodextrin (placebo for symbiotic); Behavioral: Nutritional intervention

INTERVENTIONS:
Dietary Supplement: Symbiotic — 6g sachet composition: Lactobacillus paracasei, Lactobacillus rhamnosus, Lactobacillus acidophillus, Bifidobacterium lactis and fructooligosaccharides. Each patient was instructed to consume two sachets per day, one in the morning and another before bedtime, diluted in 100 ml of filtered or boiled water at room temperature. The dietary supplement should be taken every day for 6 months.
  Arms: Symbiotic & Nutritional intervention
Dietary Supplement: Maltodextrin (placebo for symbiotic) — 6g sachet of maltodextrin, a complex carbohydrate. Each patient was instructed to consume two sachets per day, one in the morning and another before bedtime, diluted in 100 ml of filtered or boiled water at room temperature. Placebo should be taken daily for 6 months.
  Arms: Maltodextrin & Nutritional intervention
Behavioral: Nutritional intervention — Nutritional intervention consists of dietary prescription (nutritional eating plan) for healthy eating based on the Dietary Guidelines for the Brazilian Population and Clinical Manual on Food and Nutrition in HIV-infected Adults Care, both Brazil Ministry of Health guidelines, in addition to nutritional counseling for preexistent clinical conditions.

SUMMARY:
To evaluate if nutritional treatment with nutritional supplementation of dietary fiber reduces cholesterol levels and triglycerides (dyslipidemia) in patients with HIV/AIDS receiving antiretroviral therapy (HAART).

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients
* Adults (≥ 19 years old)
* On highly active antiretroviral therapy (HAART)

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Opportunistic disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Seric lipid levels | Baseline, Week 24
  Changes from baseline in total cholesterol, triglycerides, HDL-C and LDL-C.

SECONDARY OUTCOMES:
Fasting blood glucose | Baseline, Week 24
  Changes from baseline in fasting blood glucose.
Gastrointestinal symptoms | Baseline, Week 24
  Assessment of the presence of gastrointestinal symptoms (nausea and/or vomiting, dyspepsia, heartburn, diarrhea, flatulence and constipation), associated or not with antiretrorival therapy, before and after intervention to verify their effectiveness in reducing these symptoms.
Adherence to the nutritional intervention and nutritional appointments | Baseline, Week 24
  Assessment of dietary intake modification after intervention and patient's return to nutritional appointments.
Body composition | Baseline, Week 24
  Changes from baseline in total body fat percentage, percentage of fat in the trunk, percentage of fat in the arms, percentage of fat in the legs and lean body mass percentage.
Anthropometric measures | Baseline, Week 24
  Changes from baseline in weight, waist circumference, abdominal circumference, waist-to-hip ratio and Body Mass Index (BMI).

CONTACTS AND LOCATIONS:
Overall Officials: Marianne O Falco, MSc, Principal Investigator — Federal University of Goiás; Erika A Silveira, PhD, Study Director — Federal University of Goiás
Locations (1):
- Outpatient Infectoparasitary Diseases, Hospital das Clinicas, Federal University of Goiás, Goiânia, Goiás, Brazil

REFERENCES:
- [Background] Falco M, Castro Ade C, Silveira EA. [Nutritional therapy in metabolic changes in individuals with HIV/AIDS]. Rev Saude Publica. 2012 Aug;46(4):737-46. doi: 10.1590/s0034-89102012005000050. Epub 2012 Jul 10. Portuguese. PMID 22782126
- [Background] Nery MW, Martelli CM, Silveira EA, de Sousa CA, Falco Mde O, de Castro Ade C, Esper JT, Souza LC, Turchi MD. Cardiovascular risk assessment: a comparison of the Framingham, PROCAM, and DAD equations in HIV-infected persons. ScientificWorldJournal. 2013 Oct 21;2013:969281. doi: 10.1155/2013/969281. eCollection 2013. PMID 24228022
- [Derived] Santos ASEAC, Silveira EAD, Falco MO, Nery MW, Turchi MD. Effectiveness of nutritional treatment and synbiotic use on gastrointestinal symptoms reduction in HIV-infected patients: Randomized clinical trial. Clin Nutr. 2017 Jun;36(3):680-685. doi: 10.1016/j.clnu.2016.06.005. Epub 2016 Jun 23. PMID 27395330
- See also: Brazil Ministry of Health guidance on food and nutrition for patients with HIV — http://189.28.128.100/nutricao/docs/geral/manual_clinico_alimentacao_nutricao_aids_hiv.pdf